CLINICAL TRIAL: NCT00571311
Title: Parental Permission and Adolescent Assent and Decision Making in Clinical Research
Brief Title: Parental Permission and Adolescent Assent and Decision-Making in Clinical Research
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 080032; 08-CC-0032
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2018-03-12

CONDITIONS: Adolescents
Keywords: Assent; Adolescent; Informed Consent

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will evaluate how adolescents enrolled in clinical research and their parents:

* Understood the study information presented before they agreed to participate
* Made decisions about enrolling in the study
* Experienced the process of assent and consent
* Perceive the experience of participating in research

The study will determine how adolescents and their parents evaluate risk and benefit, what information they use in making their research enrollment decisions, and how these decisions are made.

In recent years the medical community and the federal government have increasingly recognized the need to conduct pediatric research. Several initiatives have resulted in an expanding number of studies that include children. With more pediatric research comes the need to ensure that protections for the rights and safety of children enrolled in research are performing well.

Adolescent patients between 13 and 18 years of age who are enrolled in a research study at the NIH involving cancer, diabetes mellitus, vaccines, obesity, bipolar disorder, and HIV, as well as healthy adolescent controls, may be eligible. One parent of each adolescent also participates.

Participants are interviewed at the NIH Clinical Center. Each interview will last about 30 minutes and consists of questions in the following areas:

* Demographics (age, sex, ethnicity, education, socioeconomic status, etc.)
* Brief medical history of the adolescent
* Experience and satisfaction with the parental permission/assent process
* Motivations for participating in clinical research
* Decision-making process
* Willingness to accept certain types and levels of hypothetical risks in a study, including those of side effects and invasive procedures
* Willingness to enroll with different chances of possible benefit
* Comparison with other activities
* General understanding of research

DETAILED DESCRIPTION:
This study aims to better understand how adolescents enrolled in clinical research and their parents understood the study information presented, made decisions about enrolling, experienced the process of assent and consent, and perceive the experience of participating in research. Interviews will be conducted with adolescents participating in clinical research and with one of their parents. Adolescents with a number of disorders including cancer, chronic diseases, bipolar disorder, obesity, and HIV, as well as healthy controls who are enrolled in NIH intramural protocols will be interviewed.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria- Adolescent:

1. Age 13 to 18.
2. Currently enrolled in clinical research.
3. Gave assent to participate in the primary study within the previous 6 months.
4. Physically and cognitively able and willing to participate in a 30-minute interview.
5. Able to understand and speak English or Spanish.

Inclusion Criteria- Parents:

1. Parent of an eligible adolescent
2. Physically and cognitively able and willing to participate in a 30 minute interview.
3. Gave permission for their child to participate in the primary study within the previous 6 months
4. Able to understand and speak English or Spanish

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 356 (Actual)
Dates: Start 2007-12-10; Study Completion 2018-03-12

CONTACTS AND LOCATIONS:
Overall Officials: Christine Grady, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Burke TM, Abramovitch R, Zlotkin S. Children's understanding of the risks and benefits associated with research. J Med Ethics. 2005 Dec;31(12):715-20. doi: 10.1136/jme.2003.003228. PMID 16319237
- [Background] Brody JL, Scherer DG, Annett RD, Pearson-Bish M. Voluntary assent in biomedical research with adolescents: a comparison of parent and adolescent views. Ethics Behav. 2003;13(1):79-95. doi: 10.1207/S15327019EB1301_10. PMID 14552306
- [Background] Brody JL, Annett RD, Scherer DG, Perryman ML, Cofrin KM. Comparisons of adolescent and parent willingness to participate in minimal and above-minimal risk pediatric asthma research protocols. J Adolesc Health. 2005 Sep;37(3):229-35. doi: 10.1016/j.jadohealth.2004.09.026. PMID 16109343